CLINICAL TRIAL: NCT03816527
Title: Selective Attention to Emotional and Alcohol-associated Cues in Patients With Alcohol Use Disorder and Healthy Participants
Brief Title: Selective Attention in Alcohol Use Disorder
Status: Withdrawn | Type: Observational
Why Stopped: study not funded / no manpower
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Other Study IDs: Emo-Dotprobe
Record Dates: First submitted 2019-01-07; First posted 2019-01-25 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AUD patients: Individuals with alcohol use disorder
- Healthy controls: Healthy controls

SUMMARY:
This study examines the selective attention to emotional- and alcohol- associated cues in alcohol- dependant and healthy participants.

DETAILED DESCRIPTION:
The planned study will investigate the selective attention to emotional and alcohol-related stimuli in alcohol-dependent patients and healthy volunteers.

background Attitudinal shifts in the implicit cognitive processing of alcohol-associated stimuli play a major role in the maintenance of addictive disorders, in the development of alcohol cravings, and ultimately in relapse. There are several experimental methods to study the selective attention to image stimuli. For preliminary studies as well as for the planned study, we opted for the so-called Dotprobe task , in which image pairs (alcohol versus neutral stimulus) are presented. The selective attention can be measured by means of reaction time differences. In addition to alcohol-related stimuli, photos of fearful and happy faces that act as emotional stimuli are also used.

In a preliminary study, the investigators were able to show that not only alcoholics, but also healthy light social drinkers, showed an initial orientation towards alcohol stimuli. The presence of such a shift in attention to alcoholic stimuli, even in healthy individuals, could be a consequence of the processing of alcoholic stimuli as emotional stimuli of increased salience compared to affectively neutral stimuli. There are still no studies that collectively examine selective attention to both emotional and alcohol-associated stimuli. While some studies have shown selective attention to fear stimuli compared to neutral stimuli only in populations with clinically relevant increased anxiety, there are also studies who were able to show that there is selective attention to evolutionarily relevant anxiety even in healthy individuals. In these non-clinical populations, this selective attention appears to be particularly prevalent in subjects with increased anxiety.

Studies using affective positive stimuli such as happy faces showed selective attention to these positive valent stimuli in healthy people compared to neutral stimuli, which was also associated with the current mood . Thus, the selective attention to cheerful faces, for example, in a positive mood was also increased. Emotional processing is relevant in the development and maintenance of addictive diseases as well as in so-called "prolonged withdrawal". Thus, during abstinence among alcoholics, increased anxiety, irritability and dysphoria, the so-called "negative emotional state of withdrawal", appear. In a functional Magnetic Resonance Imaging (fMRI) study, it was shown that when anxious faces were seen, acute alcohol abuse had anxiolytic effects. In a separate study with disgusting images on cigarette packs as an aversive fear stimuli, we found that smokers showed a shift in attention to these disgusting images was associated with relief craving and was also associated with increased anxiety, especially in heavy smokers.

Objective:

The study will compare the selective attention to emotional and alcohol-related stimuli between alcoholics and healthy people. Furthermore, their association with positive and negative mood as well as anxiety should be considered. The aim is to investigate whether alcoholic stimuli are processed the same way in healthy people, such as appetitive, emotional stimuli and whether patients' alcohol stimuli are processed like aversive, emotional stimuli.

This question is interesting both methodically and clinically. On the one hand, it would be methodologically important to interpret whether healthy alcohol-associated stimuli are appetitive or similar to affectively positive stimuli for the interpretation of studies on selective attention to alcohol stimuli and alcohol-stimulant reactivity. Clinically significant would be the identification of patients with increased selective attention to alcohol and anxiety stimuli, for whom the risk of relapse could be increased by confronting these stimuli. From these findings, therapeutic options could be derived, such as the application of exposure therapies.

Hypotheses:

1. Alcohol-dependent patients as well as healthy volunteers have a selective shift of attention to alcohol-associated versus neutral stimuli.
2. The selective attention to happy faces is associated with positive mood.
3. The selective attention to anxious faces is associated with the degree of anxiety.
4. The selective attention to anxious faces is increased in alcoholics compared to healthy controls.
5. The selective attention to happy faces is lowered in alcoholics in comparison to healthy controls.
6. Selective attention to alcohol-associated stimuli in healthy controls is associated with positive mood.
7. Selective attention to alcohol-related stimuli is associated with negative mood in alcohol-dependent patients.

Target population:

The study will examine 40 alcohol-dependent patients and 40 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing age
* Women an Men between 18 and 65 years
* Adequate ability to reach an Agreement with the Investigator, to answer oral and written questions
* Ability to consent after detailed reconnaissance
* Written informed consent
* Patients: Diagnosis of alcohol use disorder

Exclusion Criteria:

* Participants wich are unable to consent
* Severe internal, neurological ans psychiatric comorbidities
* Abstinence phenomenon (CIWA-R > 3)
* Axis I psychiatric disorder (except nicotine dependence and specific phobias within the last 12 months as well as patients with alcohol use disorder)
* Pharmacotherapy with psychoactive substances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: group 1: patients with alcohol use disorder, recruited in the Clinic of the Department of Addictive Behaviour and Addiction Medicine group 2: healthy controls, recruited from the local community
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
attentional bias to alcohol cues | at examination 1 day (single examination, no follow-up)
  measured with reaction time differences (in milliseconds) using the dotprobe-task (Vollstädt-Klein et al. 2009) [reaction time differences is not a change over time; it is measured during one experimental session]
attentional bias to emotional cues | at examination 1 day (single examination, no follow-up)
  measured with reaction time differences (in milliseconds) using the dotprobe-task (like in Vollstädt-Klein et al. 2009, but with emotional pictures) [reaction time differences is not a change over time; it is measured during one experimental session]

SECONDARY OUTCOMES:
severity of nicotine dependence | at examination 1 day (single examination, no follow-up)
  Fagerstrøm Test of Nicotine Dependence (Heatherton, Kozlowski, Frecker, & Fagerstrom, 1991)
nicotine consumption | at examination 1 day (single examination, no follow-up), retrospectively for the last 3 months
  amount of nicotine consumed during the last 3 months (like (Scheurich et al., 2005) but for nicotine instead of alcohol)
alcohol consumption | at examination 1 day (single examination, no follow-up), retrospectively for the last 3 months
  amount of alcohol consumed during the last 3 months (Scheurich et al., 2005)
severity of alcohol use disorder | at examination 1 day (single examination, no follow-up),
  Alcohol Dependence Scale, ADS (Skinner & Horn, 1984), score ranges between 0 and 47, higher score means higher severity of alcohol use disorder
habitual alcohol consumption | at examination 1 day (single examination, no follow-up), retrospectively for the last 7 days
  automated and habitual alcohol consumption during the last 7 days, measured with Craving Automated Scale for Alcohol" (CAS-A) (Vollstädt-Klein et al., 2015). 5 subscales (factors): Factor 1 ("only aware in hindsight") ranges from 0 to 35, factor 2 ("no deliberate decision") from 0 to 35, factor 3 ("contrary to intention") from 0 to 40, factor 4 ("no perception") from 0 to 20, and factor 5 ("no control") from 0 to 10. , higher score means more habitual alcohol consumption
alcohol craving | at examination 1 day (single examination, no follow-up), retrospectively for the last 7 days
  measured with Obsessive Compulsive Drinking Scale (OCDS, (Mann & Ackermann, 2000)), score ranges between 0 and 40, higher score means higher craving (obsessive-compulsive alcohol use)

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Vollstädt-Klein, Principal Investigator — ZI Mannheim
Locations (1):
- Klinik für Abhängiges Verhalten, Zentralinstitut für Seelische Gesundheit, Mannheim, Germany